CLINICAL TRIAL: NCT01683929
Title: The Effects of Oral Glucose Compared to Sweetener Drinking on Hormonal/Metabolic Responses and 24 Hour Macronutrient Consumption - A Double Blind, Cross-over Study
Brief Title: The Effects of Oral Glucose Compared to Sweetener Drinking on Hormonal/Metabolic Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: MeirMc017112CTIL
Record Dates: First submitted 2012-09-10; First posted 2012-09-12 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2014-05

CONDITIONS: Obesity
Keywords: Obesity; Overweight; Sugar consumption; Metabolic syndrome; Artificially sweetened foods and beverages
MeSH Terms: conditions — Obesity; Overweight; Metabolic Syndrome | interventions — Glucose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral glucose tolerance test (Active Comparator): The participants will consume a beverage containing 75 gram glucose During the meeting, the participants will drink the sweetened drink followed by blood work, at 0, 30, 60, 120, 180 minutes. Also, they will record their macronutrient\caloric consumption during the 24 hour following the test.
  Interventions: Other: glucose
- Artificial sweetner (Placebo Comparator): participants will consume a beverage containing 0.42 gram artificial sweetener (Aspartame) During each meeting, the participants will drink the sweetened drink followed by blood work, at 0, 30, 60, 120, 180 minutes.
  Also, they will record their macronutrient\caloric consumption during the 24 hour following the test.
  Interventions: Other: sweetner

INTERVENTIONS:
Other: glucose — The participants will report to the lab after an overnight fast. Their BMI, HR and BP will be measured. An IV catheter will be inserted into the brachial vein and the participants will rest for half an hour. Participants will drink A beverage containing 75 gram glucose (oral glucose tolerance test (OGTT / GTT) All the participants will be checked for level of: insulin, glucose, adrenalin norepinephrine, dopamine, catecholamines, cortisol, ghrelin, leptin, IGF-1 GH and other related hormones- before consuming the drink (time 0), and at 30, 60, 120, 180 minutes after.
  The participants HR & BP will be monitored throughout the examination + 1 hour after.
  In addition, the participants will be asked to complete a- "24 hr food questionnaire".
  Arms: Oral glucose tolerance test
Other: sweetner — The participants will report to the lab after an overnight fast. Their BMI, HR and BP will be measured. An IV catheter will be inserted into the brachial vein and the participants will rest for half an hour. Participants will drink A beverage containing artificial sweetened drink. All the participants will be checked for level of: insulin, glucose, adrenalin norepinephrine, dopamine, catecholamines, cortisol, ghrelin, leptin, IGF-1 GH and other related hormones- before consuming the drink (time 0), and at 30, 60, 120, 180 minutes after.
  The participants HR & BP will be monitored throughout the examination + 1 hour after.
  In addition, the participants will be asked to complete a- "24 hr food questionnaire".
  Arms: Artificial sweetner

SUMMARY:
The goal of this study is to determine the hormonal/metabolic reponse to ingestion of sugar compared to consuming artificial sweetened drink, and to evalute macronutrient consumption 24 hours post ingestion of the drinks.

We hypothesize that artificially sweetened (AS) consumption will lead to a relatively similar hormonal/metabolic responses as glucose consumption and therefore to secondary rise of caloric intake.

DETAILED DESCRIPTION:
During the last two decades, the prevalence of overweight and obesity doubled. at the same time, individuals have increasingly turned to artificially sweetened (AS) foods and beverages in an attempt to lose weight, or control it.

several studies have found that there may be a connection between artificially sweetened food and beverages consumption and paradoxical weight gain and increased incidence of metabolic syndrome. the causal relationship between AS use and weight gain haven't been proven yet.

The participants will be invited to 2 meetings in which they will consume, in a randomized double blind way:

1. A beverage containing 75 gram glucose
2. A beverage containing 0.42 gram artificially sweetener (Aspartame, similar sweetness level)

During each meeting, the participants will drink the sweetened drink followed by blood work, as done in oral glucose challenge or tolerance test (OGTT / GTT).

Also, they will record their macronutrient\caloric consumption during the 24 hour following the test.

ELIGIBILITY:
Inclusion Criteria:

* Adults, healthy, men and women, ages 25-35 years, without any chronic illnesses.

Exclusion Criteria:

* Family history of diabetes or overweight with BMI> 27
* Use of drugs who can influence the glucose metabolism (exp: glucocorticoids).

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-05; Primary Completion 2014-06 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Hormonal response | 3 hours
  All the participants will be checked for level of: insulin, glucose, adrenalin norepinephrine, dopamine, catecholamines, cortisol, ghrelin, leptin, IGF-1 GH- and other related hormones before consuming the drink (time 0), and 30, 60, 120, 180 minutes after.
  The participants will be under medical supervision throughout the examination, including HR & BP montoring, and until 1 hour after

SECONDARY OUTCOMES:
food questionnaire | 24 hours
  The participants will be receiving a- "24 hr food questionnaire" which they will fill during the day after consuming the drink followed by an interview in order to get the maximal information.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Nemet, MD, Principal Investigator — Meir Medical Center, Kfar-Saba, Israel
Locations (1):
- Meir Medical Center, Kfar Saba, Israel